CLINICAL TRIAL: NCT00620152
Title: Randomized Trial of Telephone Interventions for Pediatric Obesity in School Age Children
Brief Title: Nutrition Study for School Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Boston University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: David Ludwig, MD, PhD, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X08-01-0047 (completed); 5R01DK059240 (NIH)
Record Dates: First submitted 2008-02-19; First posted 2008-02-21 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Low glycemic load diet
  Interventions: Behavioral: 1
- 2 (Active Comparator): Low fat diet
  Interventions: Behavioral: 2

INTERVENTIONS:
Behavioral: 1 — Low glycemic load diet by telephone counseling
  Arms: 1
Behavioral: 2 — Low fat diet by telephone counseling
  Arms: 2

SUMMARY:
In this study, we evaluate whether dietary advice based on two healthy nutritional programs can be effectively delivered to families over one month by telephone. We hypothesize that among overweight school age children, a one-month telephone intervention will result in specific dietary changes consistent with the randomly assigned dietary intervention.

DETAILED DESCRIPTION:
Overweight and obesity have increasingly become problems faced by children. However, the best dietary approach for managing weight in children remains unclear and how to make dietary advice practical remains a challenge. The primary aim of the study is to evaluate the feasibility of a one-month telephone-based dietary intervention for pediatric obesity in achieving changes in the target variable (dietary glycemic load or dietary fat) of the assigned intervention. We hypothesis that among overweight school age children, a one-month telephone intervention will elicit specific dietary changes consistent with the randomly assigned prescriptions. Specifically, children counseled to reduce glycemic load will achieve a significantly greater mean reduction in glycemic load than those counseled to reduced dietary fat and, conversely, those counseled to reduce dietary fat will achieve a significantly greater mean reduction in dietary fat than those counseled to reduce glycemic load. The first ten participants enrolled will comprise a pilot study group intend to inform study design/methods and will not be included in the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 85%ile for age and sex within the last 6 months
* Living at home with a working telephone.
* Subject conversant in English
* Parent/guardian conversant and literate in English
* Family readiness to make dietary changes

Exclusion Criteria:

* Major chronic medical illness (e.g., cancer)
* Psychiatric disorder
* Obesity-associated genetic syndrome
* Current participation in another obesity-related research study or a formal weight loss program
* Family or child following a specialized diet
* Related to or living with another child study participant

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2008-04

PRIMARY OUTCOMES:
Change in diet | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Erinn Rhodes, MD, Study Director — Boston Children's Hospital; David S Ludwig, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rhodes ET, Vernacchio L, Mitchell AA, Fischer C, Giacalone P, Ludwig DS, Ebbeling CB. A telephone intervention to achieve differentiation in dietary intake: a randomized trial in paediatric primary care. Pediatr Obes. 2017 Dec;12(6):494-501. doi: 10.1111/ijpo.12171. Epub 2016 Aug 5. PMID 27492865